CLINICAL TRIAL: NCT03446183
Title: Short Term Effect of Smoking Cessation on Human Metabolism
Status: Completed | Type: Observational
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Meuhedet. Healthcare Organization (Other)
Responsible Party: Principal Investigator, Anna Aronis, Senior Lecturer, Hebrew University of Jerusalem
Other Study IDs: smoking cessation
Record Dates: First submitted 2018-02-15; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Smoking Cessation; Metabolic Syndrome
MeSH Terms: conditions — Smoking Cessation; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoking cessation prospective: Smoking cessation workshops
  Interventions: Behavioral: Smoking cessation workshops
- Smoking cessation retrospective: File review of former workshop participants
  Interventions: Behavioral: Smoking cessation workshops

INTERVENTIONS:
Behavioral: Smoking cessation workshops — All the participants took part in smoking cessation workshops. The comparison of metabolic aspects was made between the smokers and non-smokers

SUMMARY:
Investigating the short term smoking cessation on metabolism, examining of participant of smoking cessation workshops and former participants' file survey for metabolic aspects

DETAILED DESCRIPTION:
Objective: To examine metabolic aspects occurring during the first 6-12 months following smoking cessation in participants of smoking cessation workshops.

Design: A two armed study: prospective and retrospective. Prospective: Weight, BMI, waist circumference and waist: hip ratio were measured before, during and 6 months post cessation program. Retrospective: Blood test data for Blood fasting glucose (BFG) and lipid profile from the year preceding the workshops and the year after them were analyzed from participants' files. Smoking status was verified by phone conversation.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who were recruited from the smoking cessation workshops of the Meuhedet HMO (Israeli Health Services) during 2016-2017.

Exclusion Criteria:

* Candidates with benign tumors, bariatric surgeries, and endoscopic bariatric procedures before or during the study period were excluded

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers who were recruited from the smoking cessation workshops of the Meuhedet HMO (Israeli Health Services) during 2016-2017.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in weight | 6 months from baseline
  Weight in meters
Change in BMI | 6 months from baseline
  BMI in kg/m2
Change in waist and hip circumference | 6 months from baseline
  Waist and hip curcumference in centimeters
Change in Blood fasting glucose according to patient files (unspecified time points up to a year before and a year after the workshops) | up to 2 years from baseline
  BFG in mg/dl
Change in lipid profile according to patient files (unspecified time points up to a year before and a year after the workshops) | up to 2 years from baseline
  Lipid particle measurements in mg/dl

IPD SHARING:
Plan to Share IPD: No
This was not a part of Helsinki Committee approval. Anonymization of data for sharing is not expected.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT03446183/Prot_SAP_000.pdf